CLINICAL TRIAL: NCT07306650
Title: Effect of Vibrasthetic Vibration Device on Pain Reduction During Local Anesthesia in Pediatric Patients: A Randomized Clinical Study
Brief Title: Effect of Vibrasthetic Device on Pain Reduction During Local Anesthesia in Pediatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mariam Aldajani, Assistant Professor, King Abdulaziz University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 96-06-25
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Behavior Management
Keywords: Vibrasthetic; Vibration; child behavior management; local anesthesia; pediatric dentistry

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device (Experimental): This group will experience receiving a dental injection while the operator uses a vibrating device (Vibrasthetic) to vibrate the injection site.
  Interventions: Device: Vibrating device
- Manual (Active Comparator): Our study is a crossover study, so the participants will receive the dental injection while the operator manually vibrates their lip by holding the lip between their forefinger and thumb (control). The partcipants will be randomized, so phase I for the participants may be either the device or manual, and phase II will be the other method of vibration not used in phase I.
  Interventions: Procedure: Manual vibration

INTERVENTIONS:
Device: Vibrating device — Battery powered, no need to replace vibrating head of the unit (only a plastic barrier is required to cover the device), not investigated before.
  Arms: Device
Procedure: Manual vibration — The operator will hold the participant's lip between their forefinger and thumb to manually vibrate the lip and hence vibrating the injection site.
  Arms: Manual

SUMMARY:
The goal of this clinical trial is to test if children aged between 6 and 14 years who are receiving a dental injection will feel less pain by using a vibration device applied to the injection site during the injection compared to vibrating the lip using only the researcher's hands without using the vibration device. It will also test if this device makes them feel less anxious during the injection. The main question it aims to answer is:

Does using the Vibrasthetic device make dental injections more comfortable for children? Researchers will compare the effect of using this vibration device versus using their hands for manual vibration of the lip in the same child.

Participants will:

* Experience one method of vibration during their visit to the dentist (either the vibration device or manual vibration).
* then after 2 weeks they will go to the same dentist again and experience the other method of vibration.
* Receive the dental treatment they need in both visits. Participants will be asked to rate the pain they felt after the injection. This will be done by the participants choosing one of 6 pictures we will show them. Each picture explains the level of the pain they felt, and each picture has a score. We will score the pain the participants felt by looking at which picture they chose to describe their pain from the injection.

DETAILED DESCRIPTION:
Each participant will start their dental appointment by them sitting on a chair beside the dental chair and having their heart rate recorded by a pulse oximeter for baseline comfort level. They will be randomly assigned to either receive the vibration using the Vibrasthetic vibration device or by the dentist researcher manually vibrating the participant's lip during the injection. Topical anesthesia will be applied on the injection site and then they will receive the dental injection along with experiencing vibration in the area of the dental injection administered. Immediately after the injection, the participant will rate the pain intensity felt during the injection using validated Pain Scale (Wong-Baker). During the injection, a separate researcher, called the monitor, will monitor the participant's pain using the FLACC scale (Face, Legs, Activity, Cry, Consolability). Also, the monitor will record the participant's behavior using the Frankl scale, after which the participant will receiver their needed dental treatment. In the following visit, the participant will receive the other vibration method before their dental treatment with the recording of the same metrics by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-14 years
* who have previously received local anesthesia
* and whose behavior, according to the Frankl scale, was positive or definitely positive
* and the absence of systemic diseases or known allergies to local anesthetic agents

Exclusion Criteria:

* Uncooperative children
* Children with special healthcare needs
* Children with conditions affecting pain perception

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2025-12-26 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain level | Participant will record the level of pain felt immediately after receiving the injection. This usually occurs around 10 mins after the start of the appointment.
  Measured subjectively using an Arabic validated Wong-Baker Faces Pain Rating Scale by the participant choosing the picture that best describes the pain they felt. Minimum score is zero, maximum score is 10. Score of zero is the best outcome, which translates into "No hurt = no pain felt". Score of 10 is the worst outcome, which translates into "Hurts most = severe pain felt"
Pain level | Participant pain will be recorded by the investigator monitoring the participant using the scale while the patient is receiving the injection. This usually occurs around 10 mins after the start of the appointment.
  Measured objectively using Face, Legs, Activity, Cry, Consolability (FLACC) scale. The investigator monitoring the participant will record the participant's reaction while receiving the injection. Minimum score is zero, maximum score is 10. A score of zero is the best outcome, and a score of 10 is the worst outcome.
Pain level | This metric will be measured from the start of the appointment until the participant receives the injection. This will usually take around 10 minutes.
  Measured using a pulse oxymeter placed on the participant's forefinger. Pulse rate will be recorded before the participant sits on the dental chair (while they are sitting on a chair next to the dental chair) to measure baseline heart rate. Then pulse rate will be recorded again immediately by the investigator monitoring the participant after the participant receives the injection.

SECONDARY OUTCOMES:
Behavior and cooperation | This metric is measured by judging the participant's behavior, and is recorded after the injection is given. This will take around 10 mins from the start of the appointment.
  Measured using Frankl behavior scale. The investigator monitoring the participant will record the participant's behavior during and after receiving the injection. Behavior can be scored as definitely negative (--), negative (-), positive (+), or definitely positive (++). A score of (--) is the worst outcome, and a score of (++) is the best outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam B Aldajani, Principal Investigator — King Abdulaziz University
Locations (1):
- King Abdulaziz University Dental Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ching D, Finkelman M, Loo CY. Effect of the DentalVibe injection system on pain during local anesthesia injections in adolescent patients. Pediatr Dent. 2014 Jan-Feb;36(1):51-5. PMID 24717710
- [Background] Oliveira MA, Bendo CB, Ferreira MC, Paiva SM, Vale MP, Serra-Negra JM. Association between childhood dental experiences and dental fear among dental, psychology and mathematics undergraduates in Brazil. Int J Environ Res Public Health. 2012 Dec 17;9(12):4676-87. doi: 10.3390/ijerph9124676. PMID 23247225
- [Background] Kadam, N. S., Hegde, A. M., & Sharma, A. (2024). Comparative evaluation of anxiety levels in children using distraction techniques: An assessment with Venham Picture Test and pulse oximeter. Journal of Scientific Dentistry, 12(2), 95-101